CLINICAL TRIAL: NCT02333136
Title: In Vivo Raman Spectroscopy (IVRS) of Human Fingertip Capillary Beds
Brief Title: In Vivo Raman Spectroscopy of Human Capillary Beds
Acronym: IVRS
Status: Terminated | Type: Observational
Why Stopped: insufficient enrollment
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 327074-1
Record Dates: First submitted 2014-11-25; First posted 2015-01-07 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Spectrum Analysis, Raman

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IVRS studied: subjects will be monitored for changes in hematocrit based on results of in vivo raman spectroscopy scatter
  Interventions: Device: raman spectroscopy (LighTouch)

INTERVENTIONS:
Device: raman spectroscopy (LighTouch) — near infrared light will be shone upon a fingerbed capillary and light scatter measured using in vivo raman spectroscpy

SUMMARY:
The LighTouch device shines imperceptible red light into the skin and measures the light that comes back out using the method of Raman Spectroscopy. Some of this light is color shifted and some is not. Using a proprietary numerical recipe, the LighTouch device combines the signals in this remitted light and calculates hematocrit, glucose, protein and potentially other analytes. Thus the LighTouch device produces information without painful physical insult to the patient and can trend changes in these blood analytes in order to predict the need for intervention.

DETAILED DESCRIPTION:
The leading preventable cause of death for all people between 18 and 45, world-wide, military or civilian is uncontrolled internal bleeding i.e. hemorrhage. (A. Sauaia et al, J. Trauma 38, 185-193 (1995)). Internal bleeding can be very difficult to reliably detect when there is no visible external injury and the rate of blood loss is not very rapid. Two known leading indicators of blood loss are fluctuations in hematocrit and blood protein concentration. Monitoring of either of these analytes requires a blood draw and at least 3-5 minutes to obtain a single measurement. The LighTouch device shines imperceptible red light into the skin and measures the light that comes back out using the method of Raman Spectroscopy. Some of this light is color shifted and some is not. Using a proprietary numerical recipe, the LighTouch device combines the signals in this remitted light and calculates hematocrit, glucose, protein and potentially other analytes. Thus the LighTouch device produces information without painful physical insult to the patient and can trend changes in these blood analytes in order to predict the need for intervention. Previous IRB approved clinical trials over the last 10 years demonstrated useful performance for blood glucose and now the hematocrit and protein analytes are ready to be tested. Since hematocrit and protein concentrations change during hemodialysis it provides an ideal model to monitor these fluctions over time and assess the precision and accuracy of the LighTouch device for these analytes. This technique will not affect the usual dialysis treatment in any way. The subject will place one finger into the machine for exposure to the incoming light signal and sensors within the machine will detect light scatter from specfic analytes such as hematocrit. Literally hundreds of individuals have experienced the LighTouch device since 1999 and there has never been an unpleasant response or adverse outcome. The system is analagous to having a laser pointer shining on one's finger-tip. The ultimate goal of this research is to develop the device into a reliable non-invasive measure of critical blood elements that can be determined at the patient's side.

ELIGIBILITY:
Inclusion Criteria:

* adult stable on dialysis and able to consent

Exclusion Criteria:

* inability to acquire IVRS signal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stabel dialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-08; Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
correlation with actual measured hematocrit | 2 hours during dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chaiken, PhD, Principal Investigator — Syracuse University
Locations (1):
- University Dialsyis Center, Syracuse, New York, United States